CLINICAL TRIAL: NCT07310797
Title: A Randomized Controlled Trial Comparing Mirabegron and Tamsulosin for Ureteral Stone Expulsion and Clinical Symptom Improvement
Brief Title: Comparison of Mirabegron and Tamsulosin for Ureteral Stone Expulsion
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation (Other)
Responsible Party: Principal Investigator, Shu-Yu Wu, Attending Physician, Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-IRB074; TCRD-TPE-115-35 (Other Grant/Funding Number: Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation)
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Ureteral Calculi
Keywords: Mirabegron; Tamsulosin; Medical Expulsive Therapy
MeSH Terms: conditions — Ureteral Calculi | interventions — mirabegron; Tamsulosin

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of four parallel treatment groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A: Mirabegron (Experimental): Patients receive Mirabegron 50 mg daily.
  Interventions: Drug: Mirabegron
- Group B: Tamsulosin (Active Comparator): Patients receive Tamsulosin 0.4 mg daily.
  Interventions: Drug: Tamsulosin
- Group C: Combination (Experimental): Patients receive Mirabegron 50mg and Tamsulosin 0.4mg daily.
  Interventions: Drug: Mirabegron; Drug: Tamsulosin
- Group D: Standard of Care (No Intervention): Patients receive standard conservative management (symptomatic control with NSAIDs/analgesics on demand).

INTERVENTIONS:
Drug: Mirabegron — 50 mg tablet orally once daily.
  Arms: Group A: Mirabegron; Group C: Combination
Drug: Tamsulosin — 0.4 mg tablet orally once daily.
  Arms: Group B: Tamsulosin; Group C: Combination

SUMMARY:
This randomized controlled trial compares the efficacy and safety of four treatment strategies for ureteral stone expulsion: Mirabegron alone, Tamsulosin alone, a combination of both, and standard conservative care. Participants diagnosed with ureteral stones will be randomly assigned to one of these four groups. The primary objective is to evaluate the stone expulsion rate within 4 weeks. The study also assesses time to expulsion, pain intensity, analgesic use, and potential side effects.

DETAILED DESCRIPTION:
This study aims to compare the efficacy of Mirabegron, Tamsulosin, their combination, and standard conservative management in facilitating ureteral stone expulsion, as well as to evaluate their impact on clinical symptoms.

The primary objective is to analyze the differences in the stone expulsion rate within four weeks among four treatment groups:

Group A: Mirabegron 50 mg daily.

Group B: Tamsulosin 0.4 mg daily.

Group C: Combination of Mirabegron 50 mg and Tamsulosin 0.4 mg daily.

Group D: Standard of care (symptomatic control). For acute colic, Non-Steroidal Anti-Inflammatory Drugs (NSAIDs) such as Ketorolac or Diclofenac are the first-line treatment. If patients have allergies or contraindications to NSAIDs, alternative analgesics such as Tramadol or Acetaminophen will be administered.

Secondary objectives include comparing the time to stone expulsion, changes in pain intensity (assessed by Visual Analog Scale), consumption of analgesic medication, and the impact of different treatments on patient fatigue (assessed by the Fatigue Symptom Inventory, FSI).

Additionally, the study will collect and analyze adverse events occurring during the treatment period, such as palpitations, blood pressure changes, and headaches, to evaluate the safety of each intervention. The results are expected to provide comprehensive options for Medical Expulsive Therapy (MET), offering alternative non-invasive strategies for patients intolerant to traditional alpha-blockers.

ELIGIBILITY:
Inclusion Criteria:

1. Age and Sex: Adult patients aged 18 to 75 years, inclusive of both males and females.
2. Diagnosis: Unilateral ureteral stone confirmed by Computed Tomography (CT), Renal Sonography, or Kidney-Ureter-Bladder (KUB) radiography.
3. Stone Characteristics: Stone size between 4 mm and 10 mm; located in the upper (proximal), middle, or lower (distal) ureter.
4. Symptoms and Renal Function: Presence of renal colic or hematuria, with no severe renal insufficiency (eGFR > 60 mL/min/1.73m²).

Exclusion Criteria:

1. Urinary tract infection (UTI).
2. Multiple or bilateral ureteral stones.
3. Ureteral stones not visible on KUB radiography (radiolucent stones).
4. Pregnant or lactating women.
5. Severe hydronephrosis.
6. Renal insufficiency (defined as eGFR < 30 mL/min/1.73m² or Serum Creatinine > 2 mg/dL).
7. Uncontrolled hypertension or major cardiovascular disease.
8. Patients who refuse Medical Expulsive Therapy (MET).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Stone Expulsion Rate | Up to 4 weeks
  The proportion of participants with complete stone expulsion confirmed by KUB or CT scan. Successful expulsion is defined as the absence of stone fragments or the presence of clinically insignificant fragments.

SECONDARY OUTCOMES:
Time to Stone Expulsion | Up to 4 weeks
  The number of days from randomization to the confirmation of complete stone expulsion.
Change in Pain Intensity | Baseline and up to 4 weeks
  Assessed using the Visual Analog Scale (VAS), ranging from 0 (no pain) to 10 (worst possible pain).
Total Analgesic Consumption | Up to 4 weeks
  The total amount of analgesic medication (e.g., NSAIDs, Tramadol, Acetaminophen) consumed by the participant to control pain.
Change in Fatigue Symptoms | Baseline and up to 4 weeks
  Assessed using the Fatigue Symptom Inventory (FSI) to measure the intensity and interference of fatigue.
Incidence of Adverse Events | Up to 4 weeks
  Number of participants with treatment-related adverse events, such as palpitations, hypotension, dizziness, and headache.

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Yu Wu, MD, Principal Investigator — Taichung Tzu Chi Hospital
Locations (1):
- Taipei Tzu Chi Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared to protect patient confidentiality. All relevant data will be reported in the final study publication in aggregate form.